CLINICAL TRIAL: NCT04914962
Title: Wear of Enamel Antagonist to Polished Versus Glazed Zirconia Reinforced Lithium Silicate Crowns (Randomized Clinical Trial)
Brief Title: Wear of Enamel Antagonist to ZLS Crowns
Acronym: zls
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ibrahim Sameh Rady, PhD candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Wear & ZLS
Record Dates: First submitted 2021-05-29; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Wear, Tooth; Wear, Occlusal
Keywords: ZLS; crowns; occlusal wear; glass ceramic; polished vs glazed
MeSH Terms: conditions — Tooth Wear; Tooth Attrition

STUDY DESIGN:
Intervention Model Description: Patient will receive a restoration with superior function, esthetics, and excellent clinical performance
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- monolithic glazedcrowns (Active Comparator): glazed Celtra due crowns
  Interventions: Other: glazed zirconium lithium silicate
- monolithic polished crowns (Experimental): polished Celtra due crowns
  Interventions: Other: polished zirconium lithium silicate

INTERVENTIONS:
Other: glazed zirconium lithium silicate — monolithic glazed crown
  Other Names: glazed Celtra due
  Arms: monolithic glazedcrowns
Other: polished zirconium lithium silicate — monolithic polishedcrowns
  Other Names: polished Celtra due
  Arms: monolithic polished crowns

SUMMARY:
The aim of this study is to evaluate the antagonist enamel wear of two processing options of Celtra duo crowns (polished and glaze fired) restoring posterior teeth in comparison with sound enamel wear at baseline and 6 months

DETAILED DESCRIPTION:
Adhesive dental ceramics have proven to guarantee optimal esthetic results alongside satisfactory mechanical properties. Due to these qualities, today they are considered the first-choice restorative materials both for minimal restorations and for the reconstruction of severely compromised teeth. Gold alloy reconstructions preferred in the past, especially for their optimal wear properties, have been progressively substituted by these new materials.

Loss of hard tooth substance is a natural process taking place during mastication. Also, Increased wear is a common reason of failure for restorations exposed to masticatory forces. Excessive wear may be responsible for numerous problems, such as hypersensitivity, loss of occlusal contact, defects of the periodontium, reduction of masticatory efficiency, tooth migration and wrong tooth relations, weakness of masticatory muscles, and changes in the vertical and horizontal jaw relations, which may cause functional and esthetic impairments.

An optimal restorative material should provide similar characteristics to natural dental tissues. The physiological wear of enamel and dentin should represent the reference for a reasonable wear pattern of restorative materials The manufacturers tend to improve the mechanical behavior of their products leads to the progressive offer of new ceramics for daily practice. Assessment of their wear behavior and comparison through detailed tests become necessary at this point.

comparing the wear of enamel opposing polished zirconia, polished lithium disilicate crowns opposing to natural tooth. Patients were recalled after 1year and impression were recorded with opposing arch and baseline and final cast were scanned and superimposed using 3 D scanner. They found that the mean of occlusal wear of the antagonistic enamel of polished zirconia was 42.0 μm, Enamel wear against natural antagonist (control group) 34.68 μm, whereas, for Enamel wear against polished lithium disilicate crowns (group 2) 40.06 μm Enamel wear against natural antagonist (control group) 35.09 μm.

studying the quality of CAD/CAM fabricated single tooth restorations (Ten zirconia restorations were compared to 12 metal ceramic and 10 lithium disilicate counterparts). They found that were no significant differences between the studied crown systems. No difference of the gingival response among the different crown systems. Eighty percent of zirconia crowns needed no occlusal adjustment; also it showed the least amount of marginal discrepancy.

ELIGIBILITY:
Inclusion Criteria:

* Pt aged 21-60 years old, be able to read and sign the informed consent document.
* Psychologically and physically able to withstand conventional dental procedures.
* Patients needing posterior full coverage restorations
* Patients with sound natural antagonists.
* Have no active periodontal or pulpal diseases
* Able to attend punctually for preplanned visits and evaluation.

Exclusion Criteria:

* Patients with poor oral hygiene, high caries risk and uncooperative patients.
* Pregnant women.
* Psychiatric problems or unrealistic expectations.
* Lack of opposing dentition in the area of interest.
* Restored occlusal surface opposing the planned restoration.
* The presence of a removable or fixed orthodontic appliance.
* Patients with parafunctional habits.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2021-07-10 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
antagonist enamel wear | 6 months
  Intraoral digital scanner and superimposition software Mm3
  intraoral scanning of enamel antagonist to determine amount of wear in Mm3

CONTACTS AND LOCATIONS:
Overall Officials: Eman M Anwer, professor, Principal Investigator — professor of fixed prosthodontics; karim Abo Bakr Mohamed, PhD, Study Director — teacher of fixed prosthodontics

REFERENCES:
- [Background] De Angelis F, D'Arcangelo C, Maliskova N, Vanini L, Vadini M. Wear Properties of Different Additive Restorative Materials Used for Onlay/Overlay Posterior Restorations. Oper Dent. 2020 May/Jun;45(3):E156-E166. doi: 10.2341/19-115-L. Epub 2020 Feb 13. PMID 32053459
- [Background] Mehta SB, Banerji S, Millar BJ, Suarez-Feito JM. Current concepts on the management of tooth wear: part 1. Assessment, treatment planning and strategies for the prevention and the passive management of tooth wear. Br Dent J. 2012 Jan 13;212(1):17-27. doi: 10.1038/sj.bdj.2011.1099. PMID 22240686
- [Background] Dahl BL, Carlsson GE, Ekfeldt A. Occlusal wear of teeth and restorative materials. A review of classification, etiology, mechanisms of wear, and some aspects of restorative procedures. Acta Odontol Scand. 1993 Oct;51(5):299-311. doi: 10.3109/00016359309040581. PMID 8279271
- [Background] Nazirkar GS, Patil SV, Shelke PP, Mahagaonkar P. Comparative evaluation of natural enamel wear against polished yitrium tetragonal zirconia and polished lithium disilicate - An in vivo study. J Indian Prosthodont Soc. 2020 Jan-Mar;20(1):83-89. doi: 10.4103/jips.jips_218_19. Epub 2020 Jan 27. PMID 32089603
- [Background] Batson ER, Cooper LF, Duqum I, Mendonca G. Clinical outcomes of three different crown systems with CAD/CAM technology. J Prosthet Dent. 2014 Oct;112(4):770-7. doi: 10.1016/j.prosdent.2014.05.002. Epub 2014 Jun 28. PMID 24980739